CLINICAL TRIAL: NCT04053023
Title: An Open-label, Single Sequence Crossover, Drug Interaction Study to Investigate the Effect of Linerixibat (GSK2330672) on Plasma Concentrations of Obeticholic Acid and Conjugates in Healthy Participants
Brief Title: Linerixibat and Obeticholic Acid Drug Interaction Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206224
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Cholestasis
Keywords: linerixibat (GSK2330672), obeticholic acid, drug interaction, primary biliary cholangitis, pharmacokinetics
MeSH Terms: conditions — Cholestasis; Liver Cirrhosis, Biliary | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid; obeticholic acid

STUDY DESIGN:
Intervention Model Description: This will be a non-randomized study. Eligible subjects will receive OCA and OCA+linerixibat in a fixed sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants receiving obeticholic acid and linerixibat (Experimental): In Part A, participants will be administered one tablet of 10 milligrams (mg) obeticholic acid once daily continuously for 37 days (study Day 1 to study Day 37). Two tablets of 45 mg linerixibat will be administered twice daily from study Day 20 to study Day 37. 1 tablet of 45 mg linerixibat will be administered on Day 38. After evaluation of Part A, if optional part B is conducted, participants will be administered linerixibat and obeticholic acid at an alternative dosing regimen.
  Interventions: Drug: GSK2330672 (linerixibat); Drug: Obeticholic acid

INTERVENTIONS:
Drug: GSK2330672 (linerixibat) — GSK2330672 is available as a tablet with unit dose strength of 45 mg.
Drug: Obeticholic acid — Obeticholic acid is available as a tablet with a unit dose strength of 10 mg (or 5 mg dependent on evaluation of Part A).

SUMMARY:
In participants with inadequate response/intolerance to ursodeoxycholic acid (UDCA) taking obeticholic acid (OCA) who experience pruritus (due to primary biliary cholangitis [PBC], OCA, or both) the addition of linerixibat to OCA therapy may be considered following marketing approval. It is therefore important to characterize any potential effect of linerixibat on the pharmacokinetics of OCA in humans at clinically relevant dosages. Accordingly, a drug-drug interaction (DDI) study with linerixibat (potential perpetrator) and OCA (potential victim) will be conducted to inform both future clinical trials with linerixibat and the potential concomitant administration of these drugs in a clinical setting. This is a single-center, one part (with optional second part) open-label, single sequence crossover, drug interaction study to investigate the effect of linerixibat on plasma concentrations of OCA and OCA conjugates in healthy participants. Approximately 19 participants will be enrolled in part A and further 19 participants in part B (if performed) in the study and will have a phone call follow-up till 7-14 days post-last linerixibat dose.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age inclusive, at the time of signing the informed consent.
* Healthy, as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG. A participant with a clinical abnormality or laboratory parameter (i.e., outside the reference range for the population being studied), which is not specifically listed in the eligibility criteria, may be included only if the investigator agrees in consultation with the GlaxoSmithKline (GSK) medical monitor and documents in the source documentation that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or outcomes.
* Body weight > 50 kilogram (kg) and body mass index (BMI) within the range 18.5 to 32 kg per square meter (inclusive).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.
* Male and female- A female participant is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies; not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow contraceptive guidance during the treatment period and until at least 4 weeks after the last dose of study treatment. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

Exclusion Criteria:

* Any active dermatologic disorder leading to or with the potential to cause pruritus or a recent history of unexplained clinically significant itching locally or generally within the prior 3 months
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) and/or confirmed hepatocellular carcinoma or biliary cancer
* Participants with a history of cholecystectomy
* Current symptomatic cholelithiasis or inflammatory gall bladder disease
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history) clinical laboratory tests, or 12-lead ECG
* Current episode, recent history (within 1 month of screening visit), or chronic history of clinically significant diarrhea
* Lymphoma, leukaemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Any current medical condition (e.g. psychiatric disorder, senility, dementia, or other condition), clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for females and >21 units for males. One unit is equivalent to 8 gram of alcohol: a glass (approximately [~] 240 milliliter [mL]) of beer, 1 small glass (~100 mL) of wine or 1 (~25 mL) measure of spirits
* History of or regular use of tobacco- or nicotine-containing products (confirmed by smokerlyzer test) in the 3 months prior to screening.
* Administration of any IBAT inhibitor (including linerixibat) or OCA in the 3 months prior to screening
* Past or intended use of over-the-counter or prescription medication (including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless approved by the investigator in conjunction with GSK medical monitor.
* Current enrollment in a clinical trial, recent participation in a clinical trial and has received an investigational product within 30 days (or 5 half-lives of previous trial intervention, whichever is longer) before the first dose in the current study
* Exposure to more than 4 new chemical entities within 12 months before the first dose in the current study.
* Screening ALT or AST >1.5 times the upper limit of normal (ULN)
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening or within 3 months of the screening visit
* Positive serum pregnancy test at screening or positive urine pregnancy test at admission in WOCBP only
* Positive human immunodeficiency virus (HIV) antibody test
* QTc >450 millisecond (msec) on ECG performed at screening.
* Positive pre-study drug/alcohol screen or positive drug/alcohol screen at any time during the study.
* Female participants unable or unwilling to comply with specific contraception restrictions.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Unwillingness or inability to follow the procedures outlined in the protocol for the expected duration of study participation.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a data sharing agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, drug interaction study to investigate the effect of linerixibat on plasma concentrations of obeticholic acid (OCA) and OCA conjugates in healthy participants. The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 19 participants were enrolled in Part A. Part B was optional and since there was no clinical benefit seen in conducting Part B of this study, no participants were enrolled in Part B. The study was concluded following completion of Part A.
Groups:
- Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg: In Period 1, participants received OCA 10 milligram (mg), tablets, orally, once daily (afternoon dose) for 19 days (study Day 1 to Day 19). In Period 2 participants were administered OCA 10 mg, tablets, orally, once daily (afternoon dose) for 18 days (study Day 20 to Day 37) along with linerixibat 90 mg, tablets, orally, twice daily for 18.5 days (study Day 20 to the morning of Day 38). There was no washout period between Period 1 and Period 2.
- Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg: In Part B, participants were planned to receive OCA 5 mg or 10 mg, tablets, orally, once daily (evening dose) for 19 days (study Day 1 to Day 19) in Period 1; followed by OCA 10 mg, tablets, orally, once daily (evening dose) for 18 days (study Day 20 to Day 37) along with linerixibat 180 mg, tablets, orally, once daily for 18.5 days (study Day 20 to the morning of Day 38) in Period 2. There was no planned washout period between Period 1 and Period 2.
Period: Part A: Period 1 (Day 1 to Day 19)
Arm/Group | Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg | Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0
Period: Part A: Period 2 (Day 20 to Day 38)
Arm/Group | Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg | Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg
Started | 19 | 0
Completed | 18 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Part B: Period 1 (Day 1 to Day 19)
Arm/Group | Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg | Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Part B: Period 2 (Day 20 to Day 38)
Arm/Group | Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg | Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was concluded after complete analysis of Part A, there was no clinical benefit seen in conducting Part B of this study, no participants were enrolled in Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: OCA 10 mg Followed by OCA 10 mg + Linerixibat 90 mg | Part B: OCA 5mg or 10mg Followed by OCA 10mg+Linerixibat 180mg | Total
Number analyzed (Participants) | 19 | 0 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] — All Participants Population consisted of all participants who took at least 1 dose of study intervention.
  Years | 44.9 (10.28) |  | 44.9 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants] — All Participants Population consisted of all participants who took at least 1 dose of study intervention.
  Participants
    Female | 1 |  | 1
    Male | 18 |  | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — All Participants Population consisted of all participants who took at least 1 dose of study intervention.
  Participants
    Black or African American | 1 |  | 1
    White - White/Caucasian/European Heritage | 18 |  | 18

OUTCOME MEASURES:

1. Primary Outcome: Part A- Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-t]) for Total-OCA at Steady State: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of total-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Pharmacokinetic (PK) Parameters Population consisted of all participants for whom pharmacokinetic parameters were derivable.
Time Frame: Day 17: Pre-dose; Day 18: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 and 24 hours (Day 19) post-dose
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Part A: OCA 10 mg: In Part A, participants received OCA 10 mg, tablets, orally, once daily (afternoon dose) for 19 days (study Day 1 to Day 19) in Period 1.
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 2329.804 (43.54)

2. Primary Outcome: Part A- AUC(0-t) for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of total-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: Days 35 and 36: Pre-dose; Day 37: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 and 24 hours (Day 38) post-dose
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Part A: OCA 10 mg + Linerixibat 90 mg: In Part A, participants received OCA 10 mg, tablets, orally, once daily (afternoon dose) for 18 days (from study Day 20 to the Day 37) along with linerixibat 90 mg, tablets, orally, twice daily for 18.5 days (from study Day 20 to the morning of Day 38) in Period 2.
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 782.528 (55.81)

3. Primary Outcome: Part A- Area Under the Concentration-time Curve From Time 0 to 24 Hour (AUC[0-24]) for Total-OCA at Steady State: OCA Arm
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 2349.552 (43.55)

4. Primary Outcome: Part A- AUC(0-24) for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 787.007 (55.17)

5. Primary Outcome: Part A- Maximum Observed Concentration (Cmax) for Total-OCA at Steady State: OCA Arm
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 206.409 (41.18)

6. Primary Outcome: Part A- Cmax for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 83.403 (45.55)

7. Primary Outcome: Part A- Average Trough Concentration (Ctrough) for Total-OCA at Steady State: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of total-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 17, 18 and 19 has been presented.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 85.312 (53.13)

8. Primary Outcome: Part A- Average Ctrough for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of total-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 35, 36, 37 and 38 has been presented.
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 21.680 (85.11)

9. Primary Outcome: Part B- AUC(0-t) for Total-OCA at Steady State: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Groups:
- Part B: OCA 5 mg or 10 mg: In Part B, participants were planned to receive OCA 5 mg or 10 mg, tablets, orally, once daily (evening dose) for 19 days (from study Day 1 to Day 19) in Period 1.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

10. Primary Outcome: Part B- AUC(0-t) for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Groups:
- Part B: OCA 5mg or 10mg + Linerixibat 180 mg: In Part B, participants were planned to receive OCA 5 mg or 10 mg, tablets, orally, once daily (evening dose) for 18 days (from study Day 20 to the Day 37) along with linerixibat 180 mg, tablets, orally, once daily for 18.5 days (from study Day 20 to the morning of Day 38) in Period 2.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

11. Primary Outcome: Part B- AUC(0-24) for Total-OCA at Steady State: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

12. Primary Outcome: Part B- AUC(0-24) for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

13. Primary Outcome: Part B- Cmax for Total-OCA at Steady State: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

14. Primary Outcome: Part B- Cmax for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

15. Primary Outcome: Part B- Ctrough for Total-OCA at Steady State: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

16. Primary Outcome: Part B- Ctrough for Total-OCA at Steady State: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

17. Secondary Outcome: Part A- Time to Reach Maximum Observed Plasma Concentration (Tmax) for Total-OCA: OCA Arm
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours | 1.00 [0.3 to 5.0]

18. Secondary Outcome: Part A- Tmax for Total-OCA: OCA + Linerixibat Arm
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours | 3.00 [0.5 to 6.0]

19. Secondary Outcome: Part A- Assessment of Steady State Using Ctrough of Total-OCA: OCA Arm
Description: as for outcome 2
Time Frame: Day 17: Pre-dose; Day 18: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 hours and 24 hours (Day 19) post-dose
Population: PK Parameters Population.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter
  Day 17 | 92.1116 (57.86113)
  Day 18 | 95.1600 (57.50955)
  Day 19 | 102.5168 (66.65649)

20. Secondary Outcome: Part A- Assessment of Steady State Using Ctrough of Total-OCA: OCA + Linerixibat Arm
Description: as for outcome 2
Time Frame: Days 35 and 36: Pre-dose; Day 37: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 hours and 24 hours (Day 38) post-dose
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter
  Day 35 | 30.8972 (25.55139)
  Day 36 | 28.8489 (27.08479)
  Day 37 | 26.4411 (21.63264)
  Day 38 | 27.8644 (21.08848)

21. Secondary Outcome: Part A- AUC(0-t) for OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 158.337 (59.45)

22. Secondary Outcome: Part A- AUC(0-t) for OCA: OCA + Linerixibat Arm
Description: as for outcome 21
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 127.171 (53.12)

23. Secondary Outcome: Part A- AUC(0-24) for OCA: OCA Arm
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 163.701 (59.51)

24. Secondary Outcome: Part A- AUC(0-24) for OCA: OCA + Linerixibat Arm
Description: as for outcome 21
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 17
Hours * nanogram per milliliter | 130.092 (53.80)

25. Secondary Outcome: Part A- Cmax for OCA: OCA Arm
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 50.820 (71.94)

26. Secondary Outcome: Part A- Cmax for OCA: OCA + Linerixibat Arm
Description: as for outcome 21
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 35.495 (61.88)

27. Secondary Outcome: Part A- Average Ctrough for OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 17, 18 and 19 has been presented.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 2.609 (69.77)

28. Secondary Outcome: Part A- Average Ctrough for OCA: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 35, 36, 37 and 38 has been presented.
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 2.060 (83.57)

29. Secondary Outcome: Part A- Tmax for OCA: OCA Arm
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours | 0.75 [0.3 to 11.0]

30. Secondary Outcome: Part A- Tmax for OCA: OCA + Linerixibat Arm
Description: as for outcome 21
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours | 0.88 [0.5 to 12.0]

31. Secondary Outcome: Part A- AUC(0-t) for Tauro-OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of tauro-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 712.567 (61.28)

32. Secondary Outcome: Part A- AUC(0-t) for Tauro-OCA: OCA + Linerixibat Arm
Description: as for outcome 31
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 89.486 (64.85)

33. Secondary Outcome: Part A- AUC(0-24) for Tauro-OCA: OCA Arm
Description: as for outcome 31
Time Frame: as for outcome 1
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 15
Hours*nanogram per milliliter | 744.365 (68.92)

34. Secondary Outcome: Part A- AUC(0-24) for Tauro-OCA: OCA + Linerixibat Arm
Description: as for outcome 31
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 89.946 (64.50)

35. Secondary Outcome: Part A- Cmax for Tauro-OCA: OCA Arm
Description: as for outcome 31
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 62.347 (60.84)

36. Secondary Outcome: Part A- Cmax for Tauro-OCA: OCA + Linerixibat Arm
Description: as for outcome 31
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 10.224 (61.53)

37. Secondary Outcome: Part A- Average Ctrough for Tauro-OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of tauro-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 17, 18 and 19 has been presented.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 28.014 (76.45)

38. Secondary Outcome: Part A- Average Ctrough for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of tauro-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 35, 36, 37 and 38 has been presented.
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 2.600 (124.06)

39. Secondary Outcome: Part A- Tmax for Tauro-OCA: OCA Arm
Description: as for outcome 31
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours | 2.00 [0.3 to 11.0]

40. Secondary Outcome: Part A- Tmax for Tauro-OCA: OCA + Linerixibat Arm
Description: as for outcome 31
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours | 5.00 [2.0 to 9.0]

41. Secondary Outcome: Part A- AUC(0-t) for Glyco-OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of glyco-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 1741.969 (44.11)

42. Secondary Outcome: Part A- AUC(0-t) for Glyco-OCA: OCA + Linerixibat Arm
Description: as for outcome 41
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 650.683 (58.17)

43. Secondary Outcome: Part A- AUC(0-24) for Glyco-OCA: OCA Arm
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours*nanogram per milliliter | 1757.140 (44.10)

44. Secondary Outcome: Part A- AUC(0-24) for Glyco-OCA: OCA + Linerixibat Arm
Description: as for outcome 41
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours*nanogram per milliliter | 654.629 (57.45)

45. Secondary Outcome: Part A- Cmax for Glyco-OCA: OCA Arm
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 141.770 (39.46)

46. Secondary Outcome: Part A- Cmax for Glyco-OCA: OCA + Linerixibat Arm
Description: as for outcome 41
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 65.633 (50.27)

47. Secondary Outcome: Part A- Average Ctrough for Glyco-OCA: OCA Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of glyco-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 17, 18 and 19 has been presented.
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Nanogram per milliliter | 66.043 (50.72)

48. Secondary Outcome: Part A- Average Ctrough for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of glyco-OCA. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Average of Ctrough measurement from study Days 35, 36, 37 and 38 has been presented.
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Nanogram per milliliter | 19.498 (85.88)

49. Secondary Outcome: Part A- Tmax for Glyco-OCA: OCA Arm
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK Parameters Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Hours | 2.00 [0.3 to 5.0]

50. Secondary Outcome: Part A- Tmax for Glyco-OCA: OCA + Linerixibat Arm
Description: as for outcome 41
Time Frame: as for outcome 2
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Hours | 5.00 [1.0 to 6.0]

51. Secondary Outcome: Part B- Tmax for Total-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

52. Secondary Outcome: Part B- Tmax for Total-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of total-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

53. Secondary Outcome: Part B- AUC(0-t) for OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

54. Secondary Outcome: Part B- AUC(0-t) for OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

55. Secondary Outcome: Part B- AUC(0-24) for OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

56. Secondary Outcome: Part B- AUC(0-24) for OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

57. Secondary Outcome: Part B- Cmax for OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

58. Secondary Outcome: Part B- Cmax for OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

59. Secondary Outcome: Part B- Ctrough for OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

60. Secondary Outcome: Part B- Ctrough for OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

61. Secondary Outcome: Part B- Tmax for OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

62. Secondary Outcome: Part B- Tmax for OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

63. Secondary Outcome: Part B- AUC(0-t) for Tauro-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

64. Secondary Outcome: Part B- AUC(0-t) for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

65. Secondary Outcome: Part B- AUC(0-24) for Tauro-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

66. Secondary Outcome: Part B- AUC(0-24) for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

67. Secondary Outcome: Part B- Cmax for Tauro-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

68. Secondary Outcome: Part B- Cmax for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

69. Secondary Outcome: Part B- Ctrough for Tauro-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

70. Secondary Outcome: Part B- Ctrough for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

71. Secondary Outcome: Part B- Tmax for Tauro-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

72. Secondary Outcome: Part B- Tmax for Tauro-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of tauro-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

73. Secondary Outcome: Part B- AUC(0-t) for Glyco-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

74. Secondary Outcome: Part B- AUC(0-t) for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

75. Secondary Outcome: Part B- AUC(0-24) for Glyco-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

76. Secondary Outcome: Part B- AUC(0-24) for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

77. Secondary Outcome: Part B- Cmax for Glyco-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

78. Secondary Outcome: Part B- Cmax for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

79. Secondary Outcome: Part B- Ctrough for Glyco-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

80. Secondary Outcome: Part B- Ctrough for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

81. Secondary Outcome: Part B- Tmax for Glyco-OCA: OCA Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 1
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg
Number analyzed (Participants) | 0

82. Secondary Outcome: Part B- Tmax for Glyco-OCA: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of glyco-OCA.
Time Frame: as for outcome 2
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

83. Secondary Outcome: Part A- Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement. All Participants Population consisted of all participants who took at least 1 dose of study intervention.
Time Frame: Up to Day 52
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: OCA 10 mg | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 19 | 19
Participants
  Any AEs | 10 | 14
  Any SAEs | 0 | 1

84. Secondary Outcome: Part B- Number of Participants With Any AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement.
Time Frame: Up to Day 52
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

85. Secondary Outcome: Part A- Change From Baseline in PR Interval, QRS Duration, QT Interval, QT Interval Corrected Using Bazzet's Formula (QTcB), Corrected QT Interval Using Fredericia's Formula (QTcF): OCA Arm
Description: Twelve lead electrocardiograms (ECGs) were obtained to measure PR interval, QRS duration, QT interval, QTcB and QTcF. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 5 minutes. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Millisecond
  PR Interval | -3.7 (8.27)
  QRS Duration | -1.2 (4.66)
  QT Interval | -3.4 (14.56)
  QTcB Interval | 4.2 (13.31)
  QTcF Interval | 1.6 (10.43)

86. Secondary Outcome: Part A- Change From Baseline in PR Interval, QRS Duration, QT Interval, QTcB, QTcF: OCA + Linerixibat Arm
Description: Twelve lead ECGs were obtained to measure PR interval, QRS duration, QT interval, QTcB and QTcF. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 5 minutes. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Millisecond
  PR Interval | 2.5 (12.96)
  QRS Duration | -2.3 (2.97)
  QT Interval | -2.7 (13.05)
  QTcB Interval | -2.9 (13.18)
  QTcF Interval | -2.9 (9.58)

87. Secondary Outcome: Part B- Change From Baseline in PR Interval, QRS Duration, QT Interval, QTcB, QTcF
Description: Twelve lead ECGs were planned to be measured PR interval, QRS duration, QT interval, QTcB and QTcF. Twelve-lead ECGs were planned to be performed with the participant in a supine position after a rest of at least 5 minutes.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

88. Secondary Outcome: Part A- Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP): OCA Arm
Description: SBP and DBP were measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), Days 1 and 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Millimeters of mercury
  SBP: Day 1 | -0.9 (6.83)
  SBP: Day 17 | 0.5 (5.94)
  DBP: Day 1 | -4.5 (4.17)
  DBP: Day 17 | 0.1 (3.96)

89. Secondary Outcome: Part A- Change From Baseline in SBP and DBP: OCA + Linerixibat Arm
Description: as for outcome 88
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Millimeters of mercury
  SBP | -0.7 (8.48)
  DBP | 0.8 (2.98)

90. Secondary Outcome: Part A- Change From Baseline in Pulse Rate: OCA Arm
Description: Pulse rate was measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), Days 1 and 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Beats per minute
  Day 1 | 7.2 (6.54)
  Day 17 | 1.8 (7.45)

91. Secondary Outcome: Part A- Change From Baseline in Pulse Rate: OCA + Linerixibat Arm
Description: as for outcome 90
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Beats per minute | -0.3 (8.96)

92. Secondary Outcome: Part A- Change From Baseline in Respiratory Rate: OCA Arm
Description: Respiratory rate was measured in supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), Days 1 and 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Breaths per minute
  Day 1 | 0.2 (1.95)
  Day 17 | 0.4 (1.77)

93. Secondary Outcome: Part A- Change From Baseline in Respiratory Rate: OCA + Linerixibat Arm
Description: as for outcome 92
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Breaths per minute | 0.4 (2.09)

94. Secondary Outcome: Part A- Change From Baseline in Body Temperature: OCA Arm
Description: Body temperature was measured in supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1), Days 1 and 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Degrees Celsius
  Day 1 | 0.15 (0.356)
  Day 17 | 0.05 (0.336)

95. Secondary Outcome: Part A- Change From Baseline in Body Temperature: OCA + Linerixibat Arm
Description: as for outcome 94
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Degrees Celsius | 0.09 (0.327)

96. Secondary Outcome: Part B- Change From Baseline in SBP and DBP
Description: SBP and DBP were planned to be measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

97. Secondary Outcome: Part B- Change From Baseline in Pulse Rate
Description: Pulse rate was planned to be measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

98. Secondary Outcome: Part B- Change From Baseline in Respiratory Rate
Description: Respiratory rate was planned to be measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

99. Secondary Outcome: Part B- Change From Baseline in Body Temperature
Description: Body temperature was planned to be measured in a supine position after 5 minutes of rest for the participants in a quiet setting without distractions.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

100. Secondary Outcome: Part A- Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count, Leukocytes: OCA Arm
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet count and leukocytes. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
10^9 cells per liter
  Basophils | -0.002 (0.0144)
  Eosinophils | -0.013 (0.0549)
  Lymphocytes | -0.091 (0.4444)
  Monocytes | 0.033 (0.1125)
  Neutrophils | 0.064 (0.8205)
  Platelet count | 4.3 (22.85)
  Leukocytes | -0.011 (0.7760)

101. Secondary Outcome: Part A- Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count, Leukocytes: OCA + Linerixibat Arm
Description: as for outcome 100
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
10^9 cells per liter
  Basophils | 0.000 (0.0091)
  Eosinophils | 0.029 (0.0801)
  Lymphocytes | 0.169 (0.3534)
  Monocytes | 0.047 (0.0932)
  Neutrophils | 0.278 (1.2073)
  Platelet count | -4.1 (20.77)
  Leukocytes | 0.524 (1.1981)

102. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Hemoglobin: OCA Arm
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Grams per liter | 0.4 (6.33)

103. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Hemoglobin: OCA + Linerixibat Arm
Description: as for outcome 102
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Grams per liter | -0.8 (5.09)

104. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Hematocrit: OCA Arm
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Proportion of red blood cells in blood | -0.0003 (0.01614)

105. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Hematocrit: OCA + Linerixibat Arm
Description: as for outcome 104
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Proportion of red blood cells in blood | -0.0054 (0.01857)

106. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin: OCA Arm
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Picograms | -0.01 (0.624)

107. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin: OCA + Linerixibat Arm
Description: as for outcome 106
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Picograms | -0.13 (0.552)

108. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume: OCA Arm
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Femtoliter | -0.37 (1.797)

109. Secondary Outcome: Part A- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume: OCA + Linerixibat Arm
Description: as for outcome 108
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Femtoliter | -1.03 (1.972)

110. Secondary Outcome: Part A- Change From Baseline in Hematology Parameters: Erythrocytes, Reticulocytes: OCA Arm
Description: Blood samples were collected to analyze the hematology parameters: erythrocytes and reticulocytes. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
10^12 cells per liter
  Erythrocytes | 0.021 (0.1919)
  Reticulocytes | -0.0004 (0.01165)

111. Secondary Outcome: Part A- Change From Baseline in Hematology Parameters: Erythrocytes, Reticulocytes: OCA + Linerixibat Arm
Description: as for outcome 110
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
10^12 cells per liter
  Erythrocytes | 0.002 (0.2340)
  Reticulocytes | 0.0074 (0.01650)

112. Secondary Outcome: Part B- Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count, Leukocytes
Description: Blood samples were planned to be collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet count and leukocytes.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

113. Secondary Outcome: Part B- Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were planned to be collected to analyze the hematology parameter: hemoglobin.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

114. Secondary Outcome: Part B- Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were planned to be collected to analyze the hematology parameter: hematocrit.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

115. Secondary Outcome: Part B- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were planned to be collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

116. Secondary Outcome: Part B- Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were planned to be collected to analyze the hematology parameter: erythrocytes mean corpuscular volume.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

117. Secondary Outcome: Part B- Change From Baseline in Hematology Parameters: Erythrocytes, Reticulocytes
Description: Blood samples were planned to be collected to analyze the hematology parameters: erythrocytes and reticulocytes.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

118. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: Glucose, Calcium, Potassium, Sodium, Urea: OCA Arm
Description: Blood samples were collected to analyze the chemistry parameters: glucose, calcium, potassium, sodium and urea. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Millimoles per liter
  Glucose | -0.09 (0.537)
  Calcium | 0.041 (0.0891)
  Potassium | -0.02 (0.429)
  Sodium | -0.2 (2.10)
  Urea | -0.0395 (0.32717)

119. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: Glucose, Calcium, Potassium, Sodium, Urea: OCA + Linerixibat Arm
Description: as for outcome 118
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Millimoles per liter
  Glucose, n=18 | -0.44 (0.343)
  Calcium, n=18 | -0.001 (0.0506)
  Potassium, n=16: number analyzed (Participants) | 16
  Potassium, n=16 | 0.10 (0.493)
  Sodium, n=18 | -0.9 (1.89)
  Urea, n=18 | -0.1507 (0.24902)

120. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin: OCA Arm
Description: Blood samples were collected to analyze the chemistry parameters: bilirubin, creatinine and direct bilirubin. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Micromoles per liter
  Bilirubin | 0.1 (2.42)
  Creatinine | -2.2 (7.71)
  Direct Bilirubin | 0.0001 (0.88192)

121. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin: OCA + Linerixibat Arm
Description: as for outcome 120
Time Frame: Baseline (Day -1) and at Day 38
Population: as for outcome 119
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Micromoles per liter
  Bilirubin, n=18 | 1.1 (2.72)
  Creatinine, n=18 | 5.4 (6.83)
  Direct Bilirubin, n=16: number analyzed (Participants) | 16
  Direct Bilirubin, n=16 | 0.3126 (0.79317)

122. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST): OCA Arm
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP and AST. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
International units per liter
  ALT | -2.7 (4.75)
  ALP | 0.6 (5.50)
  AST | -2.2 (3.03)

123. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameters: ALT, ALP, AST: OCA + Linerixibat Arm
Description: as for outcome 122
Time Frame: Baseline (Day -1) and at Day 38
Population: as for outcome 119
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
International units per liter
  ALT, n=17: number analyzed (Participants) | 17
  ALT, n=17 | 9.4 (38.04)
  ALP, n=18 | 0.0 (9.49)
  AST, n=16: number analyzed (Participants) | 16
  AST, n=16 | -0.9 (8.50)

124. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameter: Protein: OCA Arm
Description: Blood samples were collected to analyze the chemistry parameter: protein. Baseline was considered as Day -1. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 19
Grams per liter | 1.5 (3.13)

125. Secondary Outcome: Part A- Change From Baseline in Chemistry Parameter: Protein: OCA + Linerixibat Arm
Description: as for outcome 124
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 18
Grams per liter | 0.7 (2.66)

126. Secondary Outcome: Part B- Change From Baseline in Chemistry Parameters: Glucose, Calcium, Potassium, Sodium, Urea
Description: Blood samples were planned to be collected to analyze the chemistry parameters: glucose, calcium, potassium, sodium and urea.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

127. Secondary Outcome: Part B- Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin
Description: Blood samples were planned to be collected to analyze the chemistry parameters: bilirubin, creatinine and direct bilirubin.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

128. Secondary Outcome: Part B- Change From Baseline in Chemistry Parameters: ALT, ALP, AST
Description: Blood samples were planned to be collected to analyze the chemistry parameters: ALT, ALP and AST.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

129. Secondary Outcome: Part B- Change From Baseline in Chemistry Parameter: Protein
Description: Blood samples were planned to be collected to analyze the chemistry parameter: protein.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

130. Secondary Outcome: Part A- Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline: OCA Arm
Description: Urine samples were collected from participants for urinalysis for measuring potential of hydrogen (pH) and glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocytes levels by dipstick. Abnormal urinalysis was sent for microscopic examination for cellular casts, erythrocytes, granular casts, hyaline casts, and leukocytes and were counted as cells per high-power field (cells/HPF). Baseline was considered as Day -1. Number of participants with worst case urinalysis result by microscopic examination have been presented.
Time Frame: Baseline (Day -1) and at Day 17
Population: All Participants Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: OCA 10 mg
Number analyzed (Participants) | 5
Participants
  Cellular casts: No change | 5
  Cellular casts: Increase to 1-9/HPF | 0
  Erythrocytes: No change | 4
  Erythrocytes: Increase to 1-9/HPF | 1
  Granular casts: No change | 5
  Granular casts: Increase to 1-9/HPF | 0
  Hyaline casts: No change | 5
  Hyaline casts: Increase to 1-9/HPF | 0
  Leukocytes: No change | 4
  Leukocytes: Increase to 1-9/HPF | 1

131. Secondary Outcome: Part A- Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline: OCA + Linerixibat Arm
Description: Urine samples were collected from participants for urinalysis for measuring pH and glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocytes levels by dipstick. Abnormal urinalysis was sent for microscopic examination for cellular casts, erythrocytes, granular casts, hyaline casts, and leukocytes and were counted as cells/HPF. Baseline was considered as Day -1. Number of participants with worst case urinalysis result by microscopic examination have been presented.
Time Frame: Baseline (Day -1) and at Day 38
Population: All Participants Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 1
Participants
  Cellular casts: No change | 1
  Cellular casts: Increase to 1-9/HPF | 0
  Erythrocytes: No change | 0
  Erythrocytes: Increase to 1-9/HPF | 1
  Granular casts: No change | 1
  Granular casts: Increase to 1-9/HPF | 0
  Hyaline casts: No change | 1
  Hyaline casts: Increase to 1-9/HPF | 0
  Leukocytes: No change | 1
  Leukocytes: Increase to 1-9/HPF | 0

132. Secondary Outcome: Part B- Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: Urine samples were planned to be collected from participants for urinalysis for measuring pH and glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocytes levels by dipstick. Abnormal urinalysis was planned to be sent for microscopic examination for cellular casts, erythrocytes, granular casts, hyaline casts, and leukocytes.
Time Frame: Baseline (Day -1), and up to Day 38
Population: All Participants Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5 mg or 10 mg | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0 | 0

133. Secondary Outcome: Part A- AUC(0-t) for Linerixibat: OCA + Linerixibat Arm
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of linerixibat. Pharmacokinetic parameters were analyzed using standard non-compartmental methods.
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: PK Parameters Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 19
Hours*picogram per milliliter
  Day 20, n=16: number analyzed (Participants) | 16
  Day 20, n=16 | 230.609 (153.14)
  Day 33, n=19 | 903.881 (142.27)

134. Secondary Outcome: Part A- Area Under the Concentration-time Curve From Time Zero to 12 Hours (AUC[0-12]) for Linerixibat: OCA + Linerixibat Arm
Description: as for outcome 133
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: as for outcome 133
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 17
Hours*picogram per milliliter
  Day 20, n=13: number analyzed (Participants) | 13
  Day 20, n=13 | 322.580 (121.05)
  Day 33, n=17 | 1071.982 (144.57)

135. Secondary Outcome: Part A- Cmax for Linerixibat: OCA + Linerixibat Arm
Description: as for outcome 133
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: as for outcome 133
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 19
Picogram per milliliter
  Day 20, n=17: number analyzed (Participants) | 17
  Day 20, n=17 | 56.927 (173.55)
  Day 33, n=19 | 163.624 (123.48)

136. Secondary Outcome: Part A- Tmax for Linerixibat: OCA + Linerixibat Arm
Description: as for outcome 133
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: as for outcome 133
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: OCA 10 mg + Linerixibat 90 mg
Number analyzed (Participants) | 19
Hours
  Day 20, n=17: number analyzed (Participants) | 17
  Day 20, n=17 | 3.92 [0.3 to 8.0]
  Day 33, n=19 | 5.00 [0.5 to 9.0]

137. Secondary Outcome: Part B- AUC(0-t) for Linerixibat: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of linerixibat.
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

138. Secondary Outcome: Part B- AUC(0-12) for Linerixibat: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of linerixibat.
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

139. Secondary Outcome: Part B- Cmax for Linerixibat: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of linerixibat.
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

140. Secondary Outcome: Part B- Tmax for Linerixibat: OCA + Linerixibat Arm
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of linerixibat.
Time Frame: Days 20 and 33: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post-dose
Population: PK Parameters Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: OCA 5mg or 10mg + Linerixibat 180 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected up to Day 52 in Part A
Description: All Participants Population consisted of all participants who took at least 1 dose of study intervention. Data is presented for Part A only as data was not collected for Part B since there was no clinical benefit seen in conducting Part B of this study. The study was concluded following completion of Part A.
Arm/Group | Part A: OCA 10 mg | Part A: OCA 10 mg + Linerixibat 90 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 10/19 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: OCA 10 mg (N=19) | Part A: OCA 10 mg + Linerixibat 90 mg (N=19)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: OCA 10 mg (N=19) | Part A: OCA 10 mg + Linerixibat 90 mg (N=19)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT04053023/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04053023/SAP_001.pdf